CLINICAL TRIAL: NCT04491045
Title: Randomized Control Trial on Implementation Strategies for Task-Shifting Depression Care in Vietnam
Brief Title: Implementation Strategies for Task-Shifting Depression Care Depression Care in Vietnam
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City University of New York, School of Public Health (Other)
Collaborators: Hanoi University of Public Health (Other)
Responsible Party: Principal Investigator, Victoria Ngo, Director of the Center for Innovation in Mental Health, City University of New York, School of Public Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1R01MH112630-01A1 (NIH)
Record Dates: First submitted 2020-05-13; First posted 2020-07-29 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Depression
Keywords: Behavior Activation; Problem solving therapy; Depression Treatment; Depression care integration; Implementation research; Task shifting; Collaborative care; Depression; Depressive Disorder; Behavioral Symptoms; Mood Disorders; Mental Disorders; Antidepressive Agents; Psychotropic Drugs
MeSH Terms: conditions — Depression; Depressive Disorder; Behavioral Symptoms; Mood Disorders; Mental Disorders | interventions — Organization and Administration

STUDY DESIGN:
Who Masked: Participant
Masking Description: All participants are offered depression care services at the CHS, therefore participants are not aware of the different implementation supports provided to the supervisors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Community-Engaged Learning Collaborative (CELC) (Experimental): The CELC arm is an integration of community engagement and learning collaborative approach which involves province-wide collaborative meetings for commune health stations (6 CHSs for each province) randomized into the CELC implementation condition. CELC CHSs will meet monthly initially for 3 months, followed by bi-monthly meetings for 12 months to engage in continuous quality improvement process, track implementation goals, problem solve implementation barriers, and engage in cross-site learning. This is in addition to usual implementation condition (supervision, workshops, technical assistance, and evidence-based toolkit)
  Interventions: Other: Workshop Training on Multicomponent Collaborative Care for Depression; Other: Supervision; Other: Community-Engaged Learning Collaborative
- Enhanced Supervision (ES) (Experimental): This is an evidence-based training approach which involves 6-9 months of ongoing group supervision support from psychiatric hospital mental health specialist (psychiatrist, psychiatric nurse, or psychologist) for each community health station randomized to the ES condition. Supervision approach is structured and involves observation of sessions, feedback on fidelity and quality. Supervision support will be provided biweekly initially and monthly after completion of one practice case. This is in addition to usual implementation condition (workshops, technical assistance, and evidence-based toolkit)
  Interventions: Other: Workshop Training on Multicomponent Collaborative Care for Depression; Other: Supervision
- Usual Implementation (UI) (Active Comparator): Usual Implementation (UI) Control intervention that will be enhanced usual implementation and includes hybrid training workshops on basic implementation and training supports for Multicomponent Collaborative Care for Depression program, which is an evidence-based stepped collaborative care intervention for integrating depression care into primary care settings. It consists of six components: routine screening, diagnostic assessment, psychoeducation, antidepressant medication, adherence management, behavior activation therapy.
  This implementation and training supports includes a series of online training modules, weekly webinars, and 3 one-day in-person workshops on collaborative care for depression (MCCD), limited technical assistance, and toolkit.
  Interventions: Other: Workshop Training on Multicomponent Collaborative Care for Depression

INTERVENTIONS:
Other: Workshop Training on Multicomponent Collaborative Care for Depression — Hybrid Workshop Trainings on Stepped collaborative care model for depression that involves using a team-based approach to integrating depression care components (screening, psychoeducation, Behavior Activation therapy, and antidepressant medications) into primary care settings. This integration involves task-shifting mental health tasks from mental health specialist to community providers at the commune health stations.
  Other Names: Workshop Training on Stepped collaborative care program for depression
Other: Supervision — Ongoing supervision and coaching is provided to community health providers by local mental health specialist from the provincial psychiatric hospital for 6-9 months
  Other Names: Coaching
  Arms: Community-Engaged Learning Collaborative (CELC); Enhanced Supervision (ES)
Other: Community-Engaged Learning Collaborative — The CELC group will receive support for continuous quality improvement using a province-wide learning collaborative that will meet monthly for 3 months, followed by bi-monthly meetings for 12 months.
  Other Names: Continuous Quality Improvement
  Arms: Community-Engaged Learning Collaborative (CELC)

SUMMARY:
The study is a Hybrid Implementation-Effectiveness study that will primarily test the implementation strategies on provider adoption and implementation quality in three Vietnam provinces. Secondarily, the effectiveness of the multicomponent collaborative care model for depression intervention on patient outcomes will be tested. A cluster randomized control trial design, with a mixed-methods approach, will be used to assess the effectiveness of the three implementation strategies on both organizational and provider implementation outcomes and patient effectiveness outcomes.

DETAILED DESCRIPTION:
Depression is a prevalent and debilitating mental health condition that is relatively common in almost all countries around the world, including Vietnam, and is one of the largest burdens of health. Although effective treatments exist, many with depression do not receive appropriate care. In Vietnam, numerous barriers exist to implementation of evidence-based mental health services but recently there has been growing recognition of the need to address the treatment gap. In order to close the treatment gap for depression, within the health care system, effective depression care needs to be scaled up to a wider network of community health stations that are supported by the local psychiatric hospitals. However, it is unclear what the best implementation model is for supporting depression care in primary care settings.

The aim of this project is to compare three different models of implementation support for depression care in two Vietnam provinces: 1) Supported Implementation when implementation support is provided and 2) Sustainment Phases, when study funded implementation supports are withdrawn. The providers in select community health stations (CHSs) within these two provinces) will receive training workshops and varying levels of implementation support based on the implementation models (described below) to provide depression care to their patients. The three models are : 1) Usual Implementation (UI) - a basic depression workshop, limited technical assistance to set up the program, and implementation toolkits 2) Enhanced Supervision (ES) - UI + ongoing structured supportive supervision; and 3) Community Engaged Learning Collaborative (CELC) - ES + community collaborative learning.

The three models will be evaluated based on the RE-AIM framework, which will be assessed using implementation and patient outcomes across supported implementation phase and sustainment phase. Both implementation and patient outcomes will be assessed during the sustainment phase after resources are withdrawn to evaluate the sustainability of the program. Knowledge gained from this project will be used to inform implementation of depression care services across Vietnam, and help increase access and quality of depression care.

ELIGIBILITY:
Inclusion Criteria:

Patient Participants:

* 18-65 years of age
* PHQ-9 score of 10 or above
* Planning to receive care at an eligible community health station
* Able to provide written informed consent

Provider Participants:

• General practitioners, nurses, social workers, and other qualified health care providers at a selected community health station selected by CHS Directors for depression care project.

Exclusion Criteria:

Patient Participants:

* Psychosis
* Mania
* Substance Abuse
* High suicide risk

Provider Participants: Cannot commit to full participation for the two year project period. Examples of reasons for potential barriers to commitment include leaving due to pursuit of advanced formal training at universities, anticipation of promotion or change in job status, anticipation of relocation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1382 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Provider Adoption of Project Dep and Depression Care- Count | 24 months
  Delivery of Project Dep and depression care components (Counts of depression care components delivered - # of screening, assessment, individual therapy, medication).
Provider Adoption of LIFE-DM and Depression Care - Percentage | 24 months
  Delivery of Project Dep and depression care components (% of depression care components delivered - screening, assessment, individual therapy, medication).
Change in Provider Competence Scores | 24 months
  Providers will be assessed by their supervisors for their overall competence in delivering the components of depression care every 6 months for 24 months. There are 18 items related to depression care skills (e.g., screening, psychoeducation, behavior activation, problem solving, medication management, etc.), Each item is scored on a 3 point scale from 1 to 3 (1-needs improvement, 2-satisfactory, 3-excellent). A total of 54 points can be obtained, with higher score indicating higher competence. N/A is used when a particular skill is not expected of that provider (i.e., community health workers are not expected to assess or manage medication). These ratings are conducted by supervisors at 0, 6, 12, and 24 months.
Patient Depression Scores (PHQ) Change from Baseline to 6 month | 6 months
  Patients will be assessed for depression using self-reported depression measure (PHQ). The Patient Health Questionnaire (PHQ) is a self-administered version of the PRIME-MD diagnostic instrument for common mental disorders. The PHQ-9 is the depression module, which scores each of the 9 DSM-IV criteria as "0" (not at all) to "3" (nearly every day). Total scores are used and they range from 0 to 27, with PHQ-9 scores of 5, 10, 15, and 20 represented mild, moderate, moderately severe, and severe depression, respectively.

SECONDARY OUTCOMES:
Provider Participation | 12 months
  Provider Participation in Training Activities (Count / % of workshop attendance, supervision meetings, and learning collaborative meetings).
Provider Implementation Quality | 24 months
  Supervisor Rated LIFE-DM session adherence and quality. Supervision of groups involve observation of group facilitation by supervisors, who provide adherence and quality ratings of sessions. Each item is assessed on a 4 point scale - 0 (did not do), 1 (delivered but poor), 2 (average), and 3 (excellent). The items are averaged to provide a session speciﬁc score of adherence and quality. Session adherence /quality scores are used to compute provider level adherence and quality averages. Each supervisor was expected to provide ratings for a minimum of 3 assessments out of the 12 group sessions. These session ratings are used to compute the average adherence and quality score for each provider. Higher scores indicate higher adherence and quality.
Implementation Barriers and Facilitators | 24 months
  Qualitative Interviews of Providers and Program Staff to Assess Barriers and Facilitators of Implementation
Change in Patient Functioning | 6 months
  Patient - SF-12 - Change in functioning from baseline to 6 months. The SF-12 Health Survey is a 12-item subset of the SF-36v2™ that measures the same eight domains of health (Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional, Mental Health). It is a brief, reliable measure of overall health status. Scores are calibrated so that 50 is the average score or norm. This norm-based score allows comparison among the three surveys and across the more than 19,000 studies published in the past 20 years.
Change in Patient Family Functioning | 6 months
  Patient - McMaster Family Functioning Scale - Change from baseline to 6 months. This is a 12 item scale (on a 4 point scale). the average score across items is used to determine the degree of problematic family functioning. A score of 2.00 or above indicates problematic family functioning. The higher the score, the more problematic the family member perceives the family's overall functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Ngo, PhD, Principal Investigator — City University of New York; Minh V Hoang, MD, Study Director — Hanoi University of Public Health
Locations (2):
- Vietnam (2):
  - Commune Health Stations, Bắc Giang
  - Commune Health Stations, Phú Thọ

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ngo VK, Vu TT, Vu QA, McBain R, Yu G, Nguyen NB, Mai Thi Nguyen H, Ho HT, Van Hoang M. Study protocol for type II hybrid implementation-effectiveness trial of strategies for depression care task-sharing in community health stations in Vietnam: DEP Project. BMC Public Health. 2023 Jul 28;23(1):1450. doi: 10.1186/s12889-023-16312-4. PMID 37507720